CLINICAL TRIAL: NCT04358029
Title: Cardiac Arrhythmias In Patients With Coronavirus Disease (COVID-19)
Status: Completed | Type: Observational
Sponsor: Vivek Reddy (Other)
Responsible Party: Sponsor-Investigator, Vivek Reddy, Director Cardiac Arrhythmia Service, Mount Sinai Health System, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Other Study IDs: GCO 20-0931
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: COVID 19 Cardiac; COVID 16 Arrhythmia; COVID 19 Death
Keywords: COVID 19 Cardiac; Cardiac Arrhythmias COVID

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- COVID-19 patients: Patients who have been diagnosed with COVID-19 infection at Mount Sinai Hospital
- Influenza patients: Patients who have been diagnosed with Influenza infection at Mount Sinai Hospital
- COVID-19 patients who were hospitalized with abnormal echocardiogram: Patients hospitalized for COVID-19 and who had an abnormal echocardiogram during hospitalization
- COVID-19 patients who were hospitalize with normal echocardiogram or no echocardiogram done: A matched cohort (for age, gender, troponin level, and days since hospital discharge) who did not have abnormalities on their echocardiograms (or who did not undergo echocardiogram) to ascertain that in this unusual disease, subjects did not develop echo abnormalities following hospital

SUMMARY:
The objective of the study is to estimate the frequency of cardiac arrhythmias and characterize the mode of death in patients with coronavirus disease (SARS-CoV-2; COVID-19). The study will also evaluate the long term cardiac outcomes in patients previously diagnosed with COVID-19.

This is a single-center, retrospective/ prospective registry enrolling all COVID-19 positive patients at Mount Sinai Hospital.

Cohort 1:

Retrospective chart review:

1. Patients who have been diagnosed with COVID-19 infection at Mount Sinai Hospital will be included.
2. A cohort of 1000 influenza patients will also be evaluated for purpose of comparison.

Cohort 2:

Prospective data collection of 100 patients who:

1. Were hospitalized for COVID-19 and who had an abnormal echocardiogram during hospitalization.
2. A matched cohort (for age, gender, troponin level, and days since hospital discharge) who did not have abnormalities on their echocardiograms (or who did not undergo echocardiogram) to ascertain that in this unusual disease, subjects did not develop echo abnormalities following hospital discharge.

DETAILED DESCRIPTION:
STUDY OBJECTIVE The objective of the study is to estimate the frequency of cardiac arrhythmias and characterize the mode of death in patients with the novel coronavirus disease (SARS-CoV-2; COVID-19). The study will also evaluate the long term cardiac outcomes in patients previously diagnosed with COVID-19.

INTRODUCTION, RATIONALE The novel coronavirus (SARS-CoV-2) emerged in Wuhan, China, in late 2019 and has quickly become a pandemic, significantly impacting the health and economy of the United States and the rest of the world. There are over 500,000 cases and 24,000 deaths related to COVID-19 worldwide, with an estimated mortality rate ranging from 1-8%. The United States has been impacted by this pandemic significantly with over 80,000 cases and thousands of deaths reported; these numbers will continue to worsen.

Patients infected with COVID-19 can exhibit a wide range of clinical manifestations, ranging from an asymptomatic state to mild upper respiratory symptoms (with low-grade fever) to severe disease with hypoxia and acute respiratory distress syndrome (ARDS) type lung injury. In the setting of hypoxemic respiratory failure, ground glass opacification on chest imaging is found more than 50% of the time.

COVID-19 has the potential to cause myocardial injury with at least 17% found to have an elevated troponin and 23% noted to have heart failure in a study of 191 inpatients from Wuhan, China. The prevalence of heart failure was significantly higher among non-survivors compared with survivors (52% vs. 12%). In a meta-analysis of 4 studies including a total of 341 patients, standardized mean difference of cardiac troponin I levels were significantly higher in those with severe COVID-19 related illness compared to those with non-severe disease (25.6, 95% CI 6.8-44.5). Furthermore, cases of fulminant myocarditis with cardiogenic shock have also been reported, with associated atrial and ventricular arrhythmias. In a recent report from Wuhan, China, 16.7% of hospitalized and 44.4% of ICU patients with COVID-19 had cardiac arrhythmias. Given the potential sampling bias in sicker, hospitalized patients with hypoxia and electrolyte abnormalities in the acute phase of severe illness can potentiate cardiac arrhythmias, the exact arrhythmic risk related to COVID-19 in patients with less severe illness or those who recover from the acute phase of the severe illness is currently unknown.

Furthermore, as it is currently unclear what medications may be beneficial for patients with COVID-19. Several medications eg: chloroquine, hydroxychloroquine, remdesivir, tocilizumab etc. are currently being investigated. Hydroxychloroquine is known to block Kv11.1 (HERG) and can cause drug-induced LQT. As such, these drugs are used concomitantly with other antiarrhythmic drugs such as amiodarone, Tikosyn, sotalol etc. which can be associated with QT prolongation requiring close EKG and cardiac monitoring. Improved characterization of arrhythmia burden and mechanism of death is critical, primarily in guiding the need for developing treatment strategies, additional arrhythmia monitoring and need to consider advanced prevention strategies including the role of implantable cardioverter defibrillator (ICD).

ELIGIBILITY:
Inclusion Criteria:

Cohort 1 (Retrospective):

1. Patients who have been diagnosed with COVID-19 infection at Mount Sinai Hospital will be included.
2. A cohort of 1000 influenza patients will also be evaluated for purpose of comparison.

Cohort 2 (Prospective) up to 100 patients who:

1. Were hospitalized for COVID-19 and who had an abnormal echocardiogram (~50 patients), defined as:

   1. Abnormal Left Ventricular function ( regional or global)
   2. Abnormal Right Ventricular function
   3. Pericardial effusion
   4. Diastolic dysfunction III-IV
2. A matched cohort (~50 patients, matched for age, gender, troponin level, and days since hospital discharge) who did not have abnormalities on their echocardiograms (or who did not undergo echocardiogram) to ascertain that in this unusual disease, subjects did not develop echo abnormalities following hospital discharge

Exclusion Criteria :

1. Retrospective: Individuals who have not been diagnosed with COVID-19 nor influenza.
2. Prospective: a.) Individuals who have not been diagnosed with COVID-19 b.) subjects under the age of 18 years. c.) unwilling or unable to sign consent. d.) residing in a long term care facility and unable to attend follow-up visit at MS. e.) no follow up visit conducted post-COVID hospitalization.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have been diagnosed with COVID-19 infection at Mount Sinai Hospital will be included.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Frequency of cardiac arrhythmias | 19 Months
  To characterize the frequency of cardiac arrhythmias in patients with COVID-19 infection

SECONDARY OUTCOMES:
Mode of death | 19 Months
  To characterize the mode of death in patients with COVID-19 infection
Number of recurrence of atrial arrhythmias | 19 months
  Number of recurrence of atrial arrhythmias in patients who manifested a new diagnosis atrial fibrillation or flutter while admitted with COVID-19 to evaluate long term cardiac outcomes in COVID-19 patients.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Martin Goldman, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Center for Immunization and Respiratory Diseases (NCIRD), Division of Viral Diseases. (2020, April 17). CDC: Cases of Coronavirus Disease (COVID-19) in the U.S. https://www.cdc.gov/coronavirus/2019-ncov/cases-updates/cases-in-us.html CDC_AA_refVal=https%3A%2F%2Fwww.cdc.gov%2Fcoronavirus%2F2019-ncov%2Fcases-in-us.html
- [Background] World Health Organization. (2020, April 20). WHO: Coronavirus 2019 Situation Reports. https://www.who.int/emergencies/diseases/novel-coronavirus-2019/situation-reports/
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Holshue ML, DeBolt C, Lindquist S, Lofy KH, Wiesman J, Bruce H, Spitters C, Ericson K, Wilkerson S, Tural A, Diaz G, Cohn A, Fox L, Patel A, Gerber SI, Kim L, Tong S, Lu X, Lindstrom S, Pallansch MA, Weldon WC, Biggs HM, Uyeki TM, Pillai SK; Washington State 2019-nCoV Case Investigation Team. First Case of 2019 Novel Coronavirus in the United States. N Engl J Med. 2020 Mar 5;382(10):929-936. doi: 10.1056/NEJMoa2001191. Epub 2020 Jan 31. PMID 32004427
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Lippi G, Lavie CJ, Sanchis-Gomar F. Cardiac troponin I in patients with coronavirus disease 2019 (COVID-19): Evidence from a meta-analysis. Prog Cardiovasc Dis. 2020 May-Jun;63(3):390-391. doi: 10.1016/j.pcad.2020.03.001. Epub 2020 Mar 10. No abstract available. PMID 32169400
- [Background] Hu H, Ma F, Wei X, Fang Y. Coronavirus fulminant myocarditis treated with glucocorticoid and human immunoglobulin. Eur Heart J. 2021 Jan 7;42(2):206. doi: 10.1093/eurheartj/ehaa190. No abstract available. PMID 32176300
- [Background] Liu K, Fang YY, Deng Y, Liu W, Wang MF, Ma JP, Xiao W, Wang YN, Zhong MH, Li CH, Li GC, Liu HG. Clinical characteristics of novel coronavirus cases in tertiary hospitals in Hubei Province. Chin Med J (Engl). 2020 May 5;133(9):1025-1031. doi: 10.1097/CM9.0000000000000744. PMID 32044814
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Traebert M, Dumotier B, Meister L, Hoffmann P, Dominguez-Estevez M, Suter W. Inhibition of hERG K+ currents by antimalarial drugs in stably transfected HEK293 cells. Eur J Pharmacol. 2004 Jan 19;484(1):41-8. doi: 10.1016/j.ejphar.2003.11.003. PMID 14729380
- [Result] Turagam MK, Musikantow D, Goldman ME, Bassily-Marcus A, Chu E, Shivamurthy P, Lampert J, Kawamura I, Bokhari M, Whang W, Bier BA, Malick W, Hashemi H, Miller MA, Choudry S, Pumill C, Ruiz-Maya T, Hadley M, Giustino G, Koruth JS, Langan N, Sofi A, Dukkipati SR, Halperin JL, Fuster V, Kohli-Seth R, Reddy VY. Malignant Arrhythmias in Patients With COVID-19: Incidence, Mechanisms, and Outcomes. Circ Arrhythm Electrophysiol. 2020 Nov;13(11):e008920. doi: 10.1161/CIRCEP.120.008920. Epub 2020 Oct 7. PMID 33026892